CLINICAL TRIAL: NCT03723707
Title: Enhanced Quality in Primary Care for Elders With Diabetes and Dementia
Acronym: EQUIPED-ADRD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: s18-01166; 1R21AG057291-01 (NIH)
Record Dates: First submitted 2018-10-22; First posted 2018-10-29 (Actual); Results first posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Diabetes; Dementia; Alzheimer Disease
MeSH Terms: conditions — Diabetes Mellitus; Dementia; Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (INT) (Experimental): (10 clinic sites and ~500 patients) which includes practice guidelines for clinicians, provider education, electronic health record support for quality DM-ADRD care, information about community/clinical resources, ongoing targeted provider feedback, and a panel manager (PM)
  Interventions: Behavioral: EQUIPED-ADRD Intervention
- Control (CON) (Placebo Comparator): During training the CON providers will be encouraged to do cognitive screening as well as follow the guidelines in general.
  Interventions: Behavioral: Control (CON)

INTERVENTIONS:
Behavioral: EQUIPED-ADRD Intervention — (10 clinic sites and ~500 patients) which includes practice guidelines for clinicians, provider education, electronic health record support for quality DM-ADRD care, information about community/clinical resources, ongoing targeted provider feedback, and a panel manager (PM)
  Arms: Intervention (INT)
Behavioral: Control (CON) — Will use current guidelines for primary care treatment with Diabetes and Dementia
  Arms: Control (CON)

SUMMARY:
The purpose of this study is to develop and test a care quality improvement intervention featuring use of consensus decisional guidance for the medical management of diabetes (DM) in patients with Alzheimer's disease and related dementia (ADRD) in primary care, provider (PCP) workflow enhancements supported by a panel manager(PM) for workflow support, electronic health record (EHR) decision support and feedback, and PCP collaborative learning.

ELIGIBILITY:
Inclusion Criteria:

* Patient must receive care at participating NYU FGP clinics.
* Patient must be English or Spanish speaking.
* Patient must have DM diagnosis.
* Patient must have documented cognitive impairment or an ADRD diagnosis.
* Patient must have someone who is identified as a family or friend who provides caregiving assistance.

Caregiver:

* Caregiver must have adequate knowledge of identified patient and/or participate in that member's healthcare decisions.
* Caregiver must be English or Spanish speaking.
* Caregiver must demonstrate capacity to consent to research participation.
* Caregiver must be at least 21 years old.

Exclusion Criteria:

Patient:

* Patient does not receive care at participating NYU FGP clinics.
* Patient is not 65 years and older.
* Patient is not English or Spanish speaking.
* Patient does not have DM diagnosis.
* Patient does not have documented Cognitive impairment or an ADRD diagnosis.
* Patient has severe dementia, other terminal illness with <6 months to live, and/or is hospice eligible.
* Patient does not have a caregiver.

Caregiver:

* Caregiver does not have adequate knowledge of identified patient and/or does not participate in that member's healthcare decisions.
* Caregiver is not English or Spanish speaking.
* Caregiver lacks capacity to consent to research.
* Caregiver is under 21 years old.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 355 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Chodosh, MD, MSHS, FACP, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification and publication.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Derived] Adeyemi O, Christina W, Arcila-Mesa M, Dickson VV, Ferris R, Tarpey T, Fletcher J, Blaum C, Chodosh J. Enhanced quality in primary care for elders with diabetes and dementia: Protocol for a multisite randomized controlled trial. Contemp Clin Trials. 2026 Jan;160:108165. doi: 10.1016/j.cct.2025.108165. Epub 2025 Nov 24. PMID 41297852

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention (INT) | Control (CON)
Started | 191 | 164
Completed | 68 | 78
Not Completed | 123 | 86
Not completed — Death | 32 | 32
Not completed — Admitted to long term care | 12 | 12
Not completed — No longer receiving care at NYU Langone Health | 15 | 8
Not completed — Lost to Follow-up | 40 | 22
Not completed — Discontinued after study closure | 24 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention (INT) | Control (CON) | Total
Number analyzed (Participants) | 68 | 78 | 146
Age, Continuous [Median (Standard Deviation); unit: years] | 79.5 (7.21) | 79 (7.37) | 79 (7.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 49 | 87
  Male | 30 | 29 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 29 | 53
  Not Hispanic or Latino | 44 | 49 | 93
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 6 | 12
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 13 | 14 | 27
  White | 48 | 58 | 106
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 68 | 78 | 146

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients Who Reach Consensus Target HBA1c
Description: Percentage of patients with normal HbA1c (>=7 and <=8.5) at the end of the trial after completing the 24-month Follow-up and who had reported values in their electronic health record within 6 months of study completion.
Time Frame: Up to Month 24
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Intervention (INT) | Control (CON)
Number analyzed (Participants) | 25 | 32
percentage of participants | 12 [-1.3 to 25.3] | 18.75 [4.7 to 32.8]

ADVERSE EVENTS:
Time Frame: 24 Months
Description: Adverse events were collected from notifications received from the electronic health record if the adverse event occurred within the NYU Langone Health system and the participant was enrolled in the study and from follow-up calls if the participant was reported as deceased.
Arm/Group | Intervention (INT) | Control (CON)
All-Cause Mortality (participants affected / at risk) | 33/191 | 32/164
Serious Adverse Events (participants affected / at risk) | 69/191 | 65/164
Other Adverse Events (participants affected / at risk) | 0/191 | 0/164
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention (INT) (N=191) | Control (CON) (N=164)
Abdominal pain (Gastrointestinal disorders) | 2 | 5
Acute kidney injury (Renal and urinary disorders) | 2 | 0
Agitation (Psychiatric disorders) | 0 | 2
Anemia (Blood and lymphatic system disorders) | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 1
Arterial injury (Vascular disorders) | 0 | 1
Arterial thromboembolism (Vascular disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 0 | 1
Cardiac Arrest (Cardiac disorders) | 3 | 0
Cardiac troponin increased (Investigations) | 0 | 1
Chest pain -cardiac (Cardiac disorders) | 0 | 1
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cholecystitis (Gastrointestinal disorders) | 0 | 2
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Colonic hemorrhage (Gastrointestinal disorders) | 1 | 0
Colonic Obstruction (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Death NOS (General disorders) | 28 | 20
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Delirium (Psychiatric disorders) | 2 | 2
Diarrhea (Gastrointestinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Edema limbs (General disorders) | 3 | 0
Enterocolitis infectious. (Gastrointestinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Eye infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 20 | 11
Fever (General disorders) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Gallbladder pain (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastroesophageal reflux (Gastrointestinal disorders) | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Heart Failure (Cardiac disorders) | 2 | 5
Hematoma (Vascular disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 0 | 2
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 5
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 3
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Hypothermia (General disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Injury, poisoning and procedural complications- other (Injury, poisoning and procedural complications) | 2 | 0
Intracranial hemorrhage (Nervous system disorders) | 1 | 1
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Liver Failure (Hepatobiliary disorders) | 0 | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 | 0
Lung Infection (Infections and infestations) | 4 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 3
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 1
Peripheral ischemia (Vascular disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Seizure (Nervous system disorders) | 2 | 0
Sepsis (Infections and infestations) | 1 | 1
Skin Infection (Infections and infestations) | 1 | 0
Skin Ulceration (Skin and subcutaneous tissue disorders) | 0 | 1
Social circumstances (General disorders) | 1 | 0
Stroke (Nervous system disorders) | 2 | 2
Syncope (Nervous system disorders) | 6 | 3
Thromboembolic event (Vascular disorders) | 1 | 1
Toothache (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 | 0
Upper respiratory infection (Infections and infestations) | 8 | 4
Urinary frequency (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 5
Vertigo (Ear and labyrinth disorders) | 1 | 0
Vision decreased (Eye disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Wound infection (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-20): https://cdn.clinicaltrials.gov/large-docs/07/NCT03723707/Prot_SAP_000.pdf